CLINICAL TRIAL: NCT06197620
Title: Effectiveness of Thread Embedding Acupuncture Analgesia at the EX-B2 Point at the First Lumbar Level Combined With Standard Therapy on Acute Pain and Quality of Life After Post Laparoscopic Living Donor Nephrectomy
Brief Title: Effectiveness of Thread Embedding Acupuncture Analgesia at the EX-B2 Point Combined With Standard Therapy After Laparoscopic Living Donor Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Hartono Gunarso, Medical Doctor, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-08-1375
Record Dates: First submitted 2023-11-23; First posted 2024-01-09 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Post Operative Pain, Acute; Renal Transplant Donor of Left Kidney; Quality of Life; Acupuncture Analgesia
Keywords: Laparoscopic Living Donor Nephrectomy; Post Operative Acute Pain; Quality of Life; Thread Embedding Acupuncture
MeSH Terms: conditions — Pain, Postoperative | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thread Embedding Acupuncture and Standard Therapy (Experimental): The patients are pre-operative laparoscopic living donor nephrectomy patients that receive standard analgetic drug treatment according to post-operative kidney donor transplant protocol and receive thread embedding acupuncture. All patients are also given standard therapy after surgery in the form of intravenous Paracetamol 1000 mg, 3 times a day.
  Interventions: Other: Thread embedding acupuncture and standard therapy

INTERVENTIONS:
Other: Thread embedding acupuncture and standard therapy — In the treatment, thread embedding acupuncture was performed using a needle containing polydioxanone (PDO) thread at the EX-B2 acupuncture point (12.5 mm lateral to the spinous process) at the level of the 1st lumbar vertebra with an insertion angle perpendicular to the skin surface. All patients are also given standard therapy after surgery in the form of intravenous Paracetamol 1000 mg, 3 times a day.

SUMMARY:
Kidney transplantation is the main option besides hemodialysis and continuous ambulatory peritoneal dialysis (CAPD) to prolong and improve the quality of life for patients with end-stage renal disease. The main option for obtaining organs from living donors is surgical action to remove the kidney (nephrectomy) using the laparoscopic method (laparoscopic live donor nephrectomy or LLDN). Postoperative management of LDNH in the form of intravenous paracetamol 1000 mg cannot overcome innovative pain and has drug-related risk effects.

Non-pharmacological pain management is the first line of pain management. One non-pharmacological therapy that can be an option is acupuncture. Thread embedding acupuncture (TEA) is an acupuncture method that uses certain medical threads such as catgut or polydioxanone (PDO) which are inserted into subcutaneous tissue or muscle at certain acupuncture points.

The working mechanism of TEA in treating pain is through local mechanisms in the form of releasing adenosine which binds to adenosine A1 receptors, releasing substance P, inhibiting the expression and activation of Nuclear Factor Kappa B; through a segmental mechanism in the form of a control gate mechanism; through extrasegmental mechanisms in the form of downward pain inhibition pathways; through a central mechanism in the form of release of endogenous opioids in the hypothalamus. ATB can provide a continuous stimulating effect of infiltration and acceleration of tissue regeneration, increasing anti-pain.

DETAILED DESCRIPTION:
The main outcome is to determine the effect of thread embedding acupuncture at the EX-B2 point on first lumbar on pain intensity in patients after laparoscopic living donor nephrectomy (LLDN) and to determine the effect of thread embedding acupuncture at the EX-B2 point on first lumbar on the quality of life in patients after laparoscopic living donor nephrectomy (LLDN).

The thread embedding will use Polydioxanone thread size 30G x 25,4 mm. This thread will last maximum 7 months before fully absorbed.

Pain intensity will be assessed using the VAS score 7 days before LLDN surgery (before the thread implant acupuncture procedure); and on the first, second, third, and fourteenth days after the LLDN procedure.

Quality of life scores will be measured with the Indonesian version of SF-36 questionnaire carried out seven days before LLDN surgery, on the first postoperative day, and on the fourteenth day after LLDN surgery.

The research design in this study was a case series with 6 subject only.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are prospective kidney donors who will undergo laparoscopic living donor nephrectomy (LLDN).
2. Adult patients with an age range of 21-60 years.
3. Willing to take part in this research and sign informed consent.

Exclusion Criteria:

1. The patient has a history of hypersensitive reactions to thread embedding acupuncture (TEA).
2. The patient has a history of keloids or is prone to keloid formation.
3. The patient has skin disease at the location of the TEA installation area in the back area.
4. There are abnormalities in the neurological examination of the lower extremities.
5. Have a history of spinal surgery or are scheduled to undergo spinal surgery within 7 months after the LLDN procedure.
6. There is scoliosis based on clinical examination.
7. There are other specific diagnoses that can cause secondary low back pain such as inflammatory spondylitis, spinal infection, or tumor.
8. Female patients who plan to become pregnant within 7 months after the LLDN procedure.
9. The patient has a body mass index (BMI) below 18 kg/m2
10. The patient has uncontrolled diabetes mellitus.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
Pain severity with Visual Analog Scale | 7 days before laparoscopic living donor nephrectomy and on 1st, 2nd, 14th day after laparoscopic living donor nephrectomy procedure
  Visual Analog Scale (VAS) that score 0 is no pain to 100 the worse pain A higher result means worse outcomes and lower result means better outcomes

SECONDARY OUTCOMES:
Quality of Life with Short Form 36 | 7 days before laparoscopic living donor nephrectomy, and on 1st, 2nd, and 14th day after laparoscopic living donor nephrectomy procedure
  Quality of life using Short Form 36 scoring system. It contains 8 domains such as physical function, role limitation due to physical health, role limitation due to emotional health, energy/fatigue, emotional well-being, social functioning, pain, general health. The scoring s calculated with online calculator provided by MDApp website. The result is in percentage, with higher result means better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: KEPK FKUI RSCM, Principal Investigator — Urology, University of Indonesia
Locations (1):
- Faculty of Medicine Universitas Indonesia, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: Yes